CLINICAL TRIAL: NCT06619535
Title: Sepsis As a Cause of Death Among Elderly Cancer Patients: an Updated SEER Database Analysis 2000-2021
Brief Title: Sepsis As a Cause of Death Among Elderly Cancer Patients
Status: Completed | Type: Observational
Sponsor: asmaa salama ibrahim (Other)
Responsible Party: Sponsor-Investigator, asmaa salama ibrahim, Resident physician of gastroenterology, Suez Canal University
Organization: Suez Canal University (Other)
Other Study IDs: A273
Record Dates: First submitted 2024-09-21; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Sepsis; Cancer
Keywords: sepsis; Cancer; mortality; SMR; SEER
MeSH Terms: conditions — Sepsis; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this retrospective study is to explore the association between sepsis and morality among the elderly cancer patients. Data were extracted from the Surveillance, Epidemiology and End Results( SEER) database using SEER*stat software. The study included patients aged 65 years or more who were diagnosed with cancer from 2000 to 2021. The extracted data included age, race, marital status, sex, stage, surgery, chemotherapy and radiotherapy. Multiple primary session was used to calculate the standardized Mortality ratio (SMR) as Observed/Expected with excess risk/10,000 and significance was achieved at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients
* age 65 year or more
* latency exclusion period of 0 months.

Exclusion Criteria:

- Death certificate only and autopsy only cases

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly cancer patients
Sampling Method: Probability Sample
Enrollment: 5239194 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
SMR for sepsis as a cause of death among elderly cancer patients | from Jan, 2000 till Dec, 2021
  Patients were followed up from the time of diagnosis and the risk was assessed across different time intervals: 1 year, 5 years and +10 years after cancer diagnosis from 2000 to 2021

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided